CLINICAL TRIAL: NCT04117464
Title: Efficacy of Contextual Therapies (Behavioral Activation and Acceptance and Commitment Therapy) and Cognitive Behavioral Therapy (CBT) in Group Format as a Transdiagnostic Intervention in Emotional Disorders.
Brief Title: Contextual Therapies and Cognitive Behavioral Therapy as Transdiagnostic Group Interventions for Emotional Disorders
Acronym: TRANSACTIVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oviedo (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, Concepción Fernández-Rodríguez, Professor, University of Oviedo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FPU17/01181
Record Dates: First submitted 2019-09-30; First posted 2019-10-07 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Anxiety; Depression
Keywords: anxiety; depression; behavioral activation therapy; acceptance and commitment therapy; cognitive-behavioral therapy; transdiagnostic; group therapy
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Acceptance and Commitment Therapy; Cognitive Behavioral Therapy; Control Groups

STUDY DESIGN:
Intervention Model Description: Participants are simple randomized to three experimental conditions (Behavioral activation, Acceptance and commitment therapy and Cognitive-behavior therapy) and a Wait List control group
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Behavioral activation therapy (Experimental): Behavioral activation therapy was applied following the protocol designed by Martell, Dimidjian & Herman-Dunn (2013).
  Interventions: Behavioral: Behavioral activation therapy
- Acceptance and Commitment Therapy (Experimental): Acceptance and Commitment therapy was applied following the protocol designed by Hayes, Strosahl & Wilson, (2011).
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Cognitive-Behavioral Therapy (Experimental): Cognitive-Behavioral Therapy was applied following the protocol designed by Barlow, Allen and Choate (2004).
  Interventions: Behavioral: Cognitive-Behavioral Therapy
- Wait List Group (Other): Participants at Wait List Group will be evaluated pre-post and 3, 6, 9 and 12 months follow up periods, like experimental groups.
  Interventions: Other: Wait List Group

INTERVENTIONS:
Behavioral: Behavioral activation therapy — Behavioral activation therapy administered on a group basis (maximum 6 people) over 8 weekly sessions of 90 minutes.
  Other Names: BA
  Arms: Behavioral activation therapy
Behavioral: Acceptance and Commitment Therapy — Acceptance and Commitment Therapy administered on a group basis (maximum 6 people) over 8 weekly sessions of 90 minutes.
  Other Names: ACT
  Arms: Acceptance and Commitment Therapy
Behavioral: Cognitive-Behavioral Therapy — Cognitive-Behavioral Therapy on a group basis (maximum 6 people) over 8 weekly sessions of 90 minutes.
  Other Names: CBT
  Arms: Cognitive-Behavioral Therapy
Other: Wait List Group — No psychological intervention
  Other Names: Control Group
  Arms: Wait List Group

SUMMARY:
This study aims to investigate the efficacy of three psychotherapeutic programs in group format: Acceptance and Commitment Therapy (ACT), Behavioral Activation (AC) and Transdiagnostic Cognitive Behavioral Therapy (TD-CBT), for the treatment of emotional disorders. Considering the data of the literature and the results of previous research, it is expected that this clinical investigation shows that transdiagnostic interventions that are tested (AC, ACT, TD-CBT) cause clinical changes in the post-treatment. However, it is expected that in post-treatment and in the short and medium-term follow-up, significant differences will be found between the transdiagnostic therapies examined in all outcome criteria variables; and that the greatest effectiveness and effectiveness be achieved in contextual therapies, in particular, in Behavioral Activation therapy. It is expected that the study design will allow obtaining firm evidence of the active therapeutic ingredients from the analysis of the differential efficacy of each of the psychotherapeutic programs. As a final consequence and based on the results and discussion on transdiagnostic conditions and transtherapeutic elements, it is expected to develop a unified treatment protocol (in group format -as an efficient work format and appropriate to the needs of public health services-) to be easily applied in the field of primary care. It could facilitate access to effective treatment of common mental disorders in public health services.

DETAILED DESCRIPTION:
This study aims to investigate the efficacy of three psychotherapeutic programs in group format: Acceptance and Commitment Therapy (ACT), Behavioral Activation (AC) and Transdiagnostic Cognitive Behavioral Therapy (TD-CBT), for the treatment of emotional disorders. Considering the data of the literature and the results of previous research, it is expected that this clinical investigation shows that transdiagnostic interventions that are tested (AC, ACT, TD-CBT) cause clinical changes in the post-treatment. However, it is expected that in post-treatment and in the short and medium term follow-up, significant differences will be found between the transdiagnostic therapies examined in all outcome criteria variables; and that the greatest effectiveness and effectiveness be achieved in contextual therapies, in particular, in Behavioral Activation therapy. It is expected that the study design will allow obtaining firm evidence of the active therapeutic ingredients from the analysis of the differential efficacy of each of the psychotherapeutic programs. As a final consequence and based on the results and discussion on transdiagnostic conditions and transtherapeutic elements, it is expected to develop a unified treatment protocol (in group format -as an efficient work format and appropriate to the needs of public health services-) to be easily applied in the field of primary care. It could facilitate access to effective treatment of common mental disorders in public health services.

The present investigation has as general objectives:

1. Establish the effectiveness, effectiveness and efficiency of Behavioral Activation (AC), Acceptance and Commitment (ACT) and Transdiagnostic Cognitive-Behavioral (TD-CBT) therapy applied in group format for the treatment of emotional disorders in the context of Primary Care.
2. Analyze the differential utility and adequacy of contextual transdiagnostic therapy (AC; ACT) and cognitive behavioral therapy (TD-CBT) according to clinical conditions of the disorder, characteristics of the subjects and of the therapeutic procedure and the transdiagnostic assumptions that define them.
3. Develop a unified treatment protocol for emotional disorders for implementation in primary care.

Specific objectives are:

1. Identify patterns of psychological inflexibility (experiential avoidance; activation and cognitive fusion) and cognitive biases in people with emotional disorders (anxiety and / or depression).
2. To assess the efficacy, effectiveness and efficiency of three transdiagnostic therapies (AC, ACT, and TD-CBT) applied in group format for the treatment of emotional disorders, analyzing the evolution of the outcome criteria defined in relation to emotional state and functionality of the patients assigned to each experimental treatment condition and in relation to a waiting list condition.
3. Assess the adequacy and specificity of AC, ACT and TD-CBT in the treatment of emotional disorders according to different conditions: patient's clinical state, characteristics of the context and the therapeutic procedure defined as outcome criteria variables.
4. Identify the active therapeutic ingredients of the therapies on the results of the efficacy, effectiveness and adequacy of the interventions.
5. Develop a Unified Treatment Protocol to facilitate the implementation of an efficacious and effective intervention of emotional disorders in public health institutions, especially in the context of Primary Care.
6. Maintain a website to disseminate information to general population regarding services provided in the context of this research project and to share experiences with other professionals and researchers.

The sample will be composed by patients who obtain a score that indicates clinically significant symptoms according to the Hospital Anxiety and Depression Scale (HADS, Zigmond and Snaith, 1983). All participants have to sign the informed consent after being informed about the objectives and procedure of the study.

Participants that meet inclusion criteria will be randomly assigned to the experimental and control conditions. The programs will be developed in group format (maximum 8 patients / group) and will be implemented consecutively until reaching the required sample size.

Preselected patients will be interviewed by one of the researchers. The investigator explains the objectives and procedures and then participants sign the informed consent document and answer the Hospital Anxiety and Depression Scale (HADS, Zigmond and Snaith, 1983). When the result indicates clinically significant symptoms, participants will be randomly assigned (according to the table of numbers) to one of the different conditions of the investigation: three experimental (ACT; AC; TD-TCC) and a control (WL). Next, participants will be cited for an individual evaluation session in which the study variables will be explored through clinical interview and scales. After the individual evaluation session, experimental groups will receive 8 group psychotherapy sessions specific to each condition. Then, each patient have follow ups at 3, 6, 9 and 12 months after finishing the therapeutic group.

Wait List group will be evaluated after the same period of time of the experimental groups and with the same procedure. Subsequently, participants will be offered the possibility of receiving the intervention that has been shown to be most effective and / or suitable according to their peculiarities.

Therapy was administered by two licensed clinical psychologists. In order to ensure adhesion of clinical psychologists to therapeutic protocols, the intervention sessions were audio-recorded and weekly supervision sessions by the principal investigator of study were held. In addition, regular peer-to-peer coaching and supervision meetings were held to ensure protocol adherence.

Analysis of data:

The descriptive study of the sample and a study of the equivalence of control and experimental groups (with the relevant statistics according to the type of variable) will be carried out.

The investigators will study patients evolution and compare experimental and control groups in all variables using inferential statistics and evaluate the clinical change at experimental groups. For the statistical analysis a database and the statistical program IBM SPSS will be used.

ELIGIBILITY:
Inclusion Criteria:

* Anxiety and/or depression (a score above the cutoff point in at least one of HADS subscales)
* Willingness, availability and motivation to participate in a group therapy of 8 sessions.

Exclusion Criteria:

* Being under another psychological treatment
* Physical and / or cognitive deterioration that hinders participation in the therapeutic plan.
* Serious illness that compromises patient's life and / or chronic cancer pain.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change at Depression subscale (7 items of HADS) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  frequency and intensity of depression symptoms measured by Hospital Anxiety and Depression Scale (HADS), 7 items of depression subscale
Change at Anxiety subscale (7 items of HADS) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  frequency and intensity of anxiety symptoms measured by Hospital Anxiety and Depression Scale (HADS), 7 items of anxiety subscale

SECONDARY OUTCOMES:
Change at Depression scale (BDI-IA-SCA) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  frequency and intensity of depression symptoms measured by Short form of the Beck Depression Inventory based on the cognitive-affective subscale (BDI-IA-SCA)
Change at General Anxiety scale (GAD-7) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  frequency and intensity of anxiety symptoms measured by General Anxiety Disorder Scale (GAD-7)
Change at Psychological Inflexibility scale (AAQ-II) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Change at psychological inflexibility measured by Acceptance & Action Questionnaire (AAQ-II)
Change at Behavioral activation subscale (7 items of BADS) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Behavioral activation pattern measured by 7 items of Behavioral Activation for Depression Scale (BADS) activation subscale
Change at Experiential avoidance subscale (8 items of BADS) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Experiential avoidance pattern measured by 8 items of Behavioral Activation for Depression Scale (BADS) avoidance subscale
Change at Work impairment subscale (5 items of BADS) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Degree of Work impairment measured by 5 items of Behavioral Activation for Depression Scale (BADS) work impairment subscale
Change at Social impairment (5 items of BADS) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Degree of Social impairment measured by 5 items of Behavioral Activation for Depression Scale (BADS) social impairment subscale
Change at Cognitive fusion scale (CFQ) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Cognitive fusion pattern measured by Cognitive Fusion Questionnaire (CFQ)
Change at Quality of life Scale (WHOQOL-BREF) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  General Quality of life measured by WHOQOL-BREF questionnaire
Change at Physical Health subscale (7 items of WHOQOL-BREF) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Activities of daily living, Dependence on medicinal substances and medical aids, Energy and fatigue, Mobility, Pain and discomfort, Sleep and rest and Work Capacity measured by 7 items of WHOQOL-BREF questionnaire
Change at Psychological Health subscale (6 items of WHOQOL-BREF) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Bodily image and appearance, Positive and Negative feelings, Self-esteem, Spirituality / Religion / Personal beliefs, Thinking, learning, memory and concentration, measured by 6 items of WHOQOL-BREF questionnaire
Change at Social relationships subscale (3 items of WHOQOL-BREF) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Personal relationships, Social support and Sexual activity measured by 3 items of WHOQOL-BREF questionnaire
Change at Environment subscale (8 items of WHOQOL-BREF) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Financial resources, Participation in and opportunities for recreation / leisure activities, Physical environment (pollution / noise / traffic / climate) measured by 8 items of WHOQOL-BREF questionnaire
Change at Cognitive reappraisal subscale (6 items of ERQ) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Cognitive reappraisal measured by 6 items of Emotion Regulation Questionnaire (ERQ) Reappraisal subscale
Change at Expressive suppression subscale (4 items of ERQ) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  expressive suppression measured by 4 items of Emotion Regulation Questionnaire (ERQ) suppression subscale
Change at Positive environmental reinforcement scale (EROS) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Positive environmental reinforcement perceived by the participant in recent weeks, measured by EROS (Environmental Reward Observation Scale)
Patient satisfaction scale (CSQ-8) | Post-treatment (after last session, after 8 weeks)
  Patient satisfaction measured by Client Satisfaction Questionnaire (CSQ-8)

OTHER OUTCOMES:
Change at perceived anxiety (PVAS) | At the end of session 1 (after 1 week), session 2 (after 2 weeks), session 3 (after 3 weeks), session 4 (after 4 weeks), session 5 (after 5 weeks), session 6 (after 6 weeks), session 7 (after 7 weeks) and session 8 (after 8 weeks)
  Anxiety rated by the participant by a Patients Visual analog scale (PVAS)
Change at perceived depression (PVAS) | At the end of session 1 (after 1 week), session 2 (after 2 weeks), session 3 (after 3 weeks), session 4 (after 4 weeks), session 5 (after 5 weeks), session 6 (after 6 weeks), session 7 (after 7 weeks) and session 8 (after 8 weeks)
  Depression rated by the participant by a Patients Visual analog scale (PVAS)
Change at behavioral avoidance (PVAS) | At the end of session 1 (after 1 week), session 2 (after 2 weeks), session 3 (after 3 weeks), session 4 (after 4 weeks), session 5 (after 5 weeks), session 6 (after 6 weeks), session 7 (after 7 weeks) and session 8 (after 8 weeks)
  Behavioral avoidance rated by the participant by a Patients Visual analog scale (PVAS)
Change at emotional avoidance (PVAS) | At the end of session 1 (after 1 week), session 2 (after 2 weeks), session 3 (after 3 weeks), session 4 (after 4 weeks), session 5 (after 5 weeks), session 6 (after 6 weeks), session 7 (after 7 weeks) and session 8 (after 8 weeks)
  Change at relevant activities maintenance by emotional avoidance rated by the participant by a Patients Visual analog scale (PVAS)
Change at cognitive fusion (PVAS) | At the end of session 1 (after 1 week), session 2 (after 2 weeks), session 3 (after 3 weeks), session 4 (after 4 weeks), session 5 (after 5 weeks), session 6 (after 6 weeks), session 7 (after 7 weeks) and session 8 (after 8 weeks)
  Cognitive fusion rated by the participant by a Patients Visual analog scale (PVAS)
Change at activation (PVAS) | At the end of session 1 (after 1 week), session 2 (after 2 weeks), session 3 (after 3 weeks), session 4 (after 4 weeks), session 5 (after 5 weeks), session 6 (after 6 weeks), session 7 (after 7 weeks) and session 8 (after 8 weeks)
  Activation rated by the participant by a Patients Visual analog scale (PVAS)
Self-registration techniques to asses patient adherence | At session 2 (after 2 weeks), at session 3 (after 3 weeks), at session 4 (after 4 weeks), at session 5 (after 5 weeks), at session 6 (after 6 weeks), at session 7 (after 7 weeks) and at session 8 (after 8 weeks)
  Self-registers are used during treatment sessions (after 2, 3, 4, 5, 6, 7 and 8 weeks)
Change at anxiety/irritability rated by the clinician (CVAS) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Anxiety rated by the clinician by a Clinician Visual analog scale (CVAS)
Change at depression rated by the clinician (CVAS) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Depression rated by the clinician by a Clinician Visual analog scale (CVAS)
Change at attention to the presente rated by the clinician (CVAS) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Attention to the present rated by the clinician by a Clinician Visual analog scale (CVAS)
Change at experiential avoidance rated by the clinician (CVAS) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Experiential avoidance rated by the clinician by a Clinician Visual analog scale (CVAS)
Change at emotional avoidance rated by the clinician (CVAS) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Change at relevant activities maintenance by emotional avoidance rated by the clinician by a Clinician Visual analog scale (CVAS)
Change at rumination rated by the clinician (CVAS) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Change at relevant activities maintenance by rumination rated by the clinician by a Clinician Visual analog scale (CVAS)
Change at cognitive fusion rated by the clinician (CVAS) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Change at relevant activities maintenance by cognitive fusion rated by the clinician by a Clinician Visual analog scale (CVAS)
Change at behavioral avoidance rated by the clinician (CVAS) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Behavioral avoidance rated by the clinician by a Clinician Visual analog scale (CVAS)
Change at activation rated by the clinician (CVAS) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Activation rated by the clinician by a Clinician Visual analog scale (CVAS)
Change at Avoidance of relevant activities maintained by relatives rated by the clinician (CVAS) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Avoidance of relevant activities maintained by relatives rated by the clinician by a Clinician Visual analog scale (CVAS)
Change at illness behavior maintained by relatives rated by the clinician (CVAS) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  illness Behavior maintained by relatives rated by the clinician by a Clinician Visual analog scale (CVAS)
Change at Healthy behavior promoted by relatives rated by the clinician (CVAS) | Pre-treatment, Post-treatment (after last session, after 8 weeks) and Follow ups (3, 6, 9 and 12 months)
  Healthy behavior promoted by relatives rated by the clinician by a Clinician Visual analog scale (CVAS)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication are going to be share on an official data repository (Mendeley Data)
Supporting Information: SAP, CSR

REFERENCES:
- [Derived] Fernandez-Rodriguez C, Coto-Lesmes R, Martinez-Loredo V, Gonzalez-Fernandez S, Cuesta M. Is Activation the Active Ingredient of Transdiagnostic Therapies? A Randomized Clinical Trial of Behavioral Activation, Acceptance and Commitment Therapy, and Transdiagnostic Cognitive-Behavioral Therapy for Emotional Disorders. Behav Modif. 2023 Jan;47(1):3-45. doi: 10.1177/01454455221083309. Epub 2022 Apr 15. PMID 35426318